CLINICAL TRIAL: NCT01126203
Title: Randomized Multicentre Prospective Study of Selective Laser Trabeculoplasty (SLT) vs. Argon Trabeculoplasty (ALT) in Patients With Pseudoexfoliation Glaucoma and Ocular Hypertension
Brief Title: Randomized Prospective Study of Selective Laser Trabeculoplasty (SLT) Versus Argon Trabeculoplasty (ALT) in Patients With Pseudoexfoliation Glaucoma and Ocular Hypertension
Acronym: SLT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Glaucoma Clinical Research Council (Other)
Responsible Party: Andrew CS Crichton MD, FRCS(C), University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLT1
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2010-05-24 (Estimated); Status verified 2010-05

CONDITIONS: Exfoliation Syndrome; Ocular Hypertension
Keywords: Pseudoexfoliation; Glaucoma; Ocular Hypertension; SLT; Selective Laser Trabeculoplasy (SLT); Argon Laser Trabeculoplasty (ALT)
MeSH Terms: conditions — Exfoliation Syndrome; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- selective laser trabeculoplasty (SLT) (Experimental)
  Interventions: Procedure: SLT
- Argon laser trabeculoplasty (ALT) (Experimental)
  Interventions: Procedure: ALT

INTERVENTIONS:
Procedure: SLT — All eyes will be treated using a commercially available Q-switched Nd:YAG laser (Coherent Selecta 7000, Coherent Inc., Palo Alto , CA, USA) calibrated by the manufacturer. On the day of treatment, IOP will be measured, then one drop of Apraclonidine 1% or Brimonidine 0.2% and pilocarpine 1% or 2% will be instilled. Before the patient is seated at the laser slit-lamp system a proparacaine hydrochloride drop will be instilled in the eye to be treated. A Goldmann goniolens or a Latina SLT or any other goniolens will be placed on the eye to be treated with methyl cellulose 1%. The helium-neon aiming beam is focused onto the pigmented trabecular meshwork. SLT will be performed with approximately 50 applications, a 400um spot size with energies varying from 0.8-1.2 mjoules.
  Arms: selective laser trabeculoplasty (SLT)
Procedure: ALT — All eyes will be treated using Ophthalas 532 Eyelite Laser Photocoagulator (Alcon Surgical, Dallas-Fort Worth, Texas, USA. On the day of treatment, IOP will be measured, then on the day of treatment, IOP will be measured, then one drop of Apraclonidine 1% or Brimonidine 0.2% and pilocarpine 1% will be instilled. Before the patient is seated at the laser slit-lamp system a proparacaine hydrochloride drop will be instilled in the eye to be treated. A Goldmann goniolens will be placed on the eye to be treated with methyl cellulose 1%. The aiming beam is focused onto the anterior portion of the pigmented trabecular meshwork. ALT will be performed to the superior or inferior 180 degrees with ~ 50 applications, a 50um spot size with energies varying from 400-700 mW with 0.1 second duration.
  Arms: Argon laser trabeculoplasty (ALT)

SUMMARY:
Multi-center, prospective, randomized, controlled clinical trial to compare selective laser trabeculoplasty (SLT) and Argon laser trabeculoplasty (ALT) in pseudoexfoliation glaucoma and ocular hypertension patients. IOP will be recorded, at baseline, 6 weeks, 6 months and 1 year after the laser procedure.

DETAILED DESCRIPTION:
This study derives from a clinical observation that laser treated eyed with PXF glaucoma may have a similar long-term response rates when either ALT or SLT is performed. Some authors have considered that there is a risk of IOP elevation in the immediate post laser period with ALT or SLT as a complication to be related to denser angle pigmentation (20,48). (46) No long-term analysis comparing response rates of both laser treatments in these types of patients has been done.

Primary objective is to determine which laser therapy has more IOP lowering effect as primary or adjunctive treatment in eyes diagnosed with ocular hypertension and glaucoma associated to PXF. Response rates will be compared between groups at long-term.

Secondary objective is to determine the relationship between the type of laser therapy performed and angle pigmentation, number of applications, and amount of energy used with age, number and type of medication used post laser and phakic status.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with clinical evidence of unilateral or bilateral open angle pseudoexfoliation ocular hypertension (IOP > 22mmHg) or glaucoma (Evidence on Humphrey 30-2 or Goldmann of nerve fiber layer damage) with uncontrolled IOP, over 18 years of age, and are willing to participate in the study will be included. If increased IOP is bilateral then the worst eye will be treated.

Exclusion Criteria:

* Patients will be excluded if they have evidence of any glaucoma other than pseudoexfoliative open angle, if the trabecular meshwork cannot be seen in 360 degrees, if they had previous laser therapy ALT or SLT, if they have advanced visual field defect (split fixation or a scotoma within 10 degrees fixation), taking any systemic or topical steroids, have had any previous ocular surgery (glaucoma or cataract extraction included) or laser within the previous six months, if they are monocular patients, if they have any corneal disease precluding the angle evaluation and treatment, or if they had ocular trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
IOP (Intraocular Pressure) | 1 hour, 6 weeks, 3, 6 &12 months
  The main primary outcome variable will be the intraocular pressures (IOP) at 1 hour, 6 weeks, 3, 6 & 12 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Crichton, Principal Investigator — University of Calgary
Locations (5):
- Canada (5):
  - Rockyview General Hospital Eye Clinic, Calgary, Alberta
  - St. Joseph's Health Care London Eye Clinic, London, Ontario
  - University of Ottawa Eye Institute, Ottawa, Ontario
  - Dr. C Birt, Toronto, Ontario
  - Montreal Glaucoma Institute, Montreal, Quebec

REFERENCES:
- [Derived] Rolim-de-Moura CR, Paranhos A Jr, Loutfi M, Burton D, Wormald R, Evans JR. Laser trabeculoplasty for open-angle glaucoma and ocular hypertension. Cochrane Database Syst Rev. 2022 Aug 9;8(8):CD003919. doi: 10.1002/14651858.CD003919.pub3. PMID 35943114